CLINICAL TRIAL: NCT06341452
Title: Comparison of Individualized Sodium Management Versus Standard Treatment in Hemodialysis
Acronym: SODIAH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-NaM-01-EU
Record Dates: First submitted 2023-07-30; First posted 2024-04-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease
Keywords: Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Intervention Model Description: Prospective, open, controlled, parallel, randomized, interventional, multi-center, explorative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Na zero-diffusive treatment (Other): Patients will be treated for 12 weeks sodium zero-diffusive prescription thrice weekly Hemodialysis or Hemodiafiltration sessions resulting in 36 sessions per patient.
  Interventions: Device: Hemodialysis or Hemodiafiltration either with sodium zero-diffusive treatment or standard treatment without sodium-control
- standard treatment without Na-control (Other): Patients will be treated for 12 weeks either with standard dialysate prescription thrice weekly Hemodialysis or Hemodiafiltration sessions resulting in 36 sessions per patient.
  Interventions: Device: Hemodialysis or Hemodiafiltration either with sodium zero-diffusive treatment or standard treatment without sodium-control

INTERVENTIONS:
Device: Hemodialysis or Hemodiafiltration either with sodium zero-diffusive treatment or standard treatment without sodium-control — Patients will be treated for 12 weeks thrice weekly Hemodialysis or Hemodiafiltration sessions resulting in 36 sessions per patient.

SUMMARY:
The SODIAH study is designed with the aim to assess the impact of isonatremic dialysis on interdialytic weight gain, fluid status, intradialytic hemodynamic stability, and incidence of intradialytic morbid events in dialysis patients. The study will be comparing the Na management option on the 6008 HD dialysis machines with the same machine without the Na management option turned on. Relevant performance and clinical data will be collected as well as information on patients' quality of life and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

General:

* Informed consent signed and dated by study patient and authorized physician
* Minimum age of 18 years
* The patient is legally competent and able to understand the nature, risks, meaning, and consequences of the clinical trial and can subsequently declare her/his consent for participation in the clinical trial
* Patients with a chronic kidney disease stage 5D (end stage renal disease with a glomerular filtration rate of 15 ml/min or less) on dialysis as extracorporeal renal replacement therapy.

Study-specific:

* Patients on dialysis (HD/HDF), at least 4h treatment time thrice weekly ≥ 3 months using a standard dialysate with a prescribed sodium concentration of 136 mmol/L
* Anuric patients (<300mL/d; 1 measurement within last 4 weeks)
* Patient fulfils one of the four following criteria:

interdialytic weight gain over 4% of dry weight (mean value during run-in period) OR pre-dialytic systolic blood pressure over 180 mmHg (mean value during run-in period) OR intradialytic morbid events (hypotension, hypertension, cramps, headache) in at least three sessions during run-in period OR volume overload according to BCM (FO ≥2.5 L pre-dialysis or relative FO pre-dialysis ≥15% for men and ≥13% for women; one measurement during run-in period)

- Patients with a diffusive Na load of at least 1 mmoL/(L TBW) or 0.06g NaCl/(L TBW) (mean value during the run-in period).

Exclusion Criteria:

General:

* Any conditions which could interfere with the patient's ability to comply with the study
* Patient is not able to give informed consent according to European Medical Device Regulation and corresponding national regulations
* In case of female patients: pregnancy (pregnancy test will be conducted at start and end of study with female patients aged ≤55 years) or lactation period
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study

Study-specific:

* Patients treated with individualized sodium management over the last 3 months
* Severe hypoalbuminemia (≤30 g/L; 1 measurement within last 4 weeks)
* Hypernatremia (pre-dialytic plasma sodium concentration ≥145mmol/L; 1 measurement within last 4 weeks)
* Uncontrolled diabetic patients with glycated hemoglobin (HbA1C) >8%; 1 measurement within last 4 weeks
* Impossible reliable measurement of the different compartments by bioimpedance due to lower limb amputation or wearing of a unipolar pacemaker or metallic prostheses
* Life expectancy less than 6 months
* ONLINEplus HF treatments/hemofiltration treatments
* Single-needle treatments
* Dry weight < 40kg
* Active or chronic infections (HIV, SARS-CoV-2, HBV, HCV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Interdialytic weight gain | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on interdialytic weight gain will be analyzed in kg and % of dry weight
Intradialytic hemodynamic stability | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on intradialytic hemodynamic stability will be analyzed based on frequency of intradialytic hypotensive episodes
Intradialytic hemodynamic stability | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on intradialytic hemodynamic stability will be analyzed based on frequency of intradialytic hypertensive episodes
Intradialytic morbid events | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on the frequency of intradialytic morbid events will be analyzed
Fluid status | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on fluid status will be analyzed with regard to overhydration (L)
Fluid status | 12 weeks after start of study
  Evaluation of the impact of sodium zero-diffusive dialysis on fluid status will be analyzed with regard to dry weight (kg)

SECONDARY OUTCOMES:
PRO: Thirst feeling | 12 weeks after start of study
  Evaluation of thirst feeling will be assessed via the Dialysis Thirst Inventory
PRO: Thirst feeling | 12 weeks after start of study
  Evaluation of thirst feeling will be assessed via the Xerostomia Inventory
PRO: Fatigue | 12 weeks after start of study
  Evaluation of fatigue will be assessed via the CONVINCE Dialysis Fatigue Scale (CFDS-10)
PRO: Hypotensive episodes | 12 weeks after start of study
  Evaluation of hypotensive episodes will be assessed via the CONVINCE intradialytic symptoms (IDS) Scale - hypotensive episodes items
PRO: HRQOL | 12 weeks after start of study
  Evaluation of health related quality of life (HRQOL) will be assessed using the validated Kidney Disease Quality of Life (KDQOL) survey KDQOL-36
PRO: Health status | 12 weeks after start of study
  Evaluation of health status will be assessed via the validated EQ-5D-5L survey by EuroQol group

CONTACTS AND LOCATIONS:
Overall Officials: Martin Jirovec, Dr., Principal Investigator — Fresenius Medical Care - DS, s.r.o., Marianske Lazne; Czech Republic; Björn Meijers, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen Leuven, Leuven, Belgium; Maria Jesus Izquierdo Ortiz, Dr., Principal Investigator — Burgos University Hospital, Burgos, Spain
Locations (1):
- Fresenius Medical Care- DS, s.r.o., Mariánské Lázně, Czechia

IPD SHARING:
Plan to Share IPD: No